CLINICAL TRIAL: NCT01941173
Title: A Prospective Study of Short Infusion of Ziv-Aflibercept in Combination With FOLFIRI in Patients With Metastatic Colorectal Cancer
Brief Title: Short-Infusion Ziv-aflibercept in Treating Patients With Metastatic Colorectal Cancer Receiving Combination Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13294; NCI-2013-01727 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13294 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — aflibercept; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ziv-aflibercept, FOLFIRI) (Experimental): Patients receive ziv-aflibercept IV over 15-30 minutes followed by FOLFIFRI chemotherapy comprising leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Drug: leucovorin calcium; Drug: irinotecan hydrochloride; Drug: fluorouracil

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
This pilot clinical trial studies short-infusion ziv-aflibercept in treating patients with metastatic colorectal cancer receiving combination chemotherapy. Ziv-aflibercept may stop the growth of colorectal cancer by blocking blood flow to the tumor. Giving the drug over a shorter infusion time may result in improved efficiency and patient satisfaction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of a shorter infusion of 30 minutes and 15 minutes of standard dose ziv-aflibercept when combined with FOLFIRI (folinic acid [leucovorin calcium], fluorouracil, and irinotecan [irinotecan hydrochloride]) in patients with metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. Describe the institutional safety experience with this combination using Common Terminology Criteria for Adverse Events (CTCAE) version 4 for toxicity grading.

OUTLINE:

Patients receive ziv-aflibercept intravenously (IV) over 15-30 minutes followed by FOLFIFRI chemotherapy comprising leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer are eligible for this study; colorectal cancer should have been previously confirmed by pathology or cytology; to be eligible for this protocol, patients should be receiving ziv-aflibercept plus FOLFIRI as a standard treatment prior to enrolling on this trial; the number and type of therapy administered prior to enrollment will not affect the ability to enroll on this study
* Patients should have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients should have an expected life expectancy of 12 weeks or longer
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* To be eligible for this study, patients should already be receiving a standard dose of ziv-aflibercept intravenously over 60 minutes in combination with FOLFIRI chemotherapy every 2 weeks without evidence of progressive disease; treatment on this study can start as early as two weeks from last "off protocol" ziv-aflibercept plus FOLFIRI cycle, granted treatment parameters have been met
* Total bilirubin < 1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 ULN unless patient has metastatic disease to the liver in which case < 5 ULN will be allowed
* Serum creatinine < 1.5 ULN
* Urine protein/creatinine ration (UPCR) =< 1 or total urinary protein of < 1 gm/24 hours in the event the UPCR > 1
* Systolic blood pressure < 155 mm mercury and diastolic blood pressure < 100 mm mercury documented on two separate occasions at least 24 hours apart
* Platelet counts >= 75,000/mm^3
* Neutrophil count >= 1500/mm^3
* Hemoglobin >= 9 gm/dl; anemia can be corrected with transfusion to allow eligibility prior to enrollment
* Hematological tests can be repeated to assess eligibility
* No unresolved grade 2 or above non-hematological toxicities, with the exception of alopecia or neuropathy
* All subjects must have the ability to understand and the willingness to sign a written consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness such as congestive heart failure, respiratory distress, and including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy with the exception of study drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ziv-aflibercept
* Patients should be at least 2 weeks from their last dose of ziv-aflibercept when they receive their first dose of study treatment
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this study
* Patients with other active malignancies are ineligible for this study with the exception of non-melanoma skin cancer that is amenable to excision, cervical carcinoma in situ, hormone sensitive prostate cancer, or prostate cancer with no measurable disease (watchful waiting)
* History of arterial thrombotic events within 1 year prior to enrollment on study
* Surgical intervention within 4 weeks prior to study initiation and no open wounds
* Clinically significant bleeding; clinically significant bleeding is defined as gastrointestinal bleeding requiring a blood transfusion, bleeding manifesting as melena, or blood per rectum estimated to exceed 2 tablespoons within 4 weeks prior to enrollment; hemoptysis associated with blood loss of more than 1/2 tablespoon per day is also considered significant; physician judgment will be used to estimate presence or lack of significant clinical bleeding
* History of bowel perforation
* History of intracranial bleeding
* History of reversible posterior leukoencephalopathy syndrome (RPLS)
* History of active fistula
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of a shorter infusion time, determined by rate of greater or equal to grade 2 hypersensitivity reactions as graded according to CTCAE version 4.0 | Up to 30 days after last study treatment
  All hypersensitivity grades will be collected (including grade 1). Upon completion of the study, toxicity will be summarized and tabulated.

SECONDARY OUTCOMES:
Incidence of grade 3 and above toxicities, graded according to CTCAE version 4.0 | Up to 30 days after last study treatment
  Upon completion of the study, toxicity will be summarized and tabulated.

OTHER OUTCOMES:
Time on protocol therapy | Up to 30 days after last study treatment
  Summarized using range, median, and quartiles of time and total courses.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope- South Pasadena Cancer Center, South Pasadena, California